CLINICAL TRIAL: NCT05154630
Title: Phase I Clinical Trial Evaluating the Tolerability and Pharmacokinetics of TQB2858 Injection in Subjects With Advanced Malignancies
Brief Title: Study on Tolerability and Pharmacokinetics of TQB2858 Injection in Subjects With Advanced Malignant Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor has decided to terminate this study based on the current clinical research status of dual antibody drugs and full communication with the investigators.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-I-05
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Advanced Cancer; Advanced Soft-tissue Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 injection (Experimental): Participants will receive 3 mg/60 mg/600 mg/1200 mg/1800 mg single dose of TQB2858 injection on Day 1, iv (injection of vein), once every three weeks.
  Interventions: Drug: TQB2858 injection

INTERVENTIONS:
Drug: TQB2858 injection — TQB2858 is a Programmed cell death 1 ligand 1 (PD-L1)/transforming growth factor-β(TGF-β) double antibody.

SUMMARY:
This study is divided into two phases: dose escalation and cohort expansion. The dose escalation stage aims to evaluate the tolerability, pharmacokinetic characteristics and safety of TQB2858 injection in subjects with advanced malignant tumors. The cohort expansion phase aims to evaluate the initial efficacy and safety of TQB2858 injection in patients with soft tissue sarcoma, and to explore treatment-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Phase I (dose-escalation phase).

  a) Patients with advanced malignant solid/hematologic tumors who have a histologically and/or cytologically confirmed diagnosis and who have failed standard therapy or lack effective therapies.
* Phase II (cohort expansion phase).

  1. Unresectable, recurrent or metastatic adenoid soft tissue sarcoma diagnosed by histology.
  2. Previously received anti-vascular targeted drug therapy
  3. Have at least one measurable lesion Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Age: 18 to 70 years old;
* The Eastern Cooperative Oncology Group (ECOG) score: 0 to 1;
* The expected survival period is ≥3 months;
* Normal function of major organs
* Women of childbearing age should agree to use effective contraceptive measures during the study period and 6 months after the end of the study, and have a negative serum or urine pregnancy test within 7 days before enrollment in the study; men should agree to use effective contraception during the study period and after the end of the study period 6 Effective contraceptive measures must be used within one month.
* Patients voluntarily enroll in this study, sign an informed consent form and comply well.

Exclusion Criteria:

* Combined diseases and medical history:

  1. Have presented with or currently have concurrent other malignancies within 2 years.
  2. Unresolved toxic reactions due to any prior treatment above Common Terminology Criteria for Adverse Events(CTCAE) grade 1, excluding alopecia, peripheral sensory nerve disorders.
  3. Major surgical treatment or significant traumatic injury within 28 days prior to the start of study treatment.
  4. Long-term untreated wounds or fractures.
  5. An arterial/venous thrombotic event within 6 months, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism.
  6. Persons with a history of psychotropic substance abuse who are unable to abstain or have a mental disorder.
  7. Subjects with any severe and/or uncontrollable disease, including:
* Tumor-related symptoms and treatment:

  1. Have received surgery, chemotherapy, radiotherapy or other anti-cancer therapy within 4 weeks prior to the start of study treatment.
  2. Treatment with proprietary Chinese medicines with clear antitumor indications in the National Medical Products Administration (NMPA)-approved drug formulary within 2 weeks prior to the start of study treatment.
  3. Prior receipt of immune dual anti-treatment drugs against the same target of TQB2858 injection.
  4. Uncontrolled pleural effusions, pericardial effusions, or ascites that still require repeated drainage (in the judgment of the investigator);
  5. Brain metastases with less than 4 weeks of stable symptom control after discontinuation of dehydrating agents and steroids.
* Research and treatment related:

  1. History of live attenuated vaccination within 28 days prior to the start of study treatment.
  2. Prior history of severe allergy to macromolecular drugs or allergy to known components of TQB2858 injection.
  3. Active autoimmune disease requiring systemic therapy that occurred within 2 years prior to the start of study treatment.
  4. Diagnosis of immunodeficiency or being treated with systemic glucocorticoids or any other form of immunosuppressive therapy.
* Participation in other clinical trials of antineoplastic drugs within 4 weeks prior to enrollment.
* Subjects who, in the judgment of the investigator, have a concomitant illness that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or for whom other reasons are deemed to exist for ineligibility for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 48 weeks
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD.
Overall response rate (ORR) | up to 48 weeks
  ORR refers to the percentage of complete response (CR) or partial response (PR) subjects determined by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or iRECIST (CR and PR under iRECIST criteria can occur after imaging disease progression).

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to 48 weeks
  DCR refers to the percentage of subjects with CR, PR, or stable disease (SD) of 6 weeks or more as determined by RECIST 1.1 or iRECIST (CR, PR, SD under iRECIST criteria can occur after imaging disease progression).
Overall survival (OS) | Baseline up to die
  OS is defined as the time from enrollment to death from any cause.
Progression-Free Survival (PFS) | up to 48 weeks
  PFS will be defined as median number of months from the date of randomization until the first documented sign of disease progression or death due to any causes, whichever occurs first.
Duration of Response (DOR) | up to 48 weeks
  DOR will be defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan